CLINICAL TRIAL: NCT03687515
Title: Efficacy and Safety of Budesonide Inhalation Suspension Via Transnasal Nebulization Compared With Budesonide Aqueous Nasal Spray and Oral Steroids for the Treatment of Chronic Rhinosinusitis With Polyposis.
Brief Title: Efficacy and Safety of Budesonide Inhalation Suspension for the Treatment of Chronic Rhinosinusitis With Polyposis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-BIS
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Chronic Rhinosinusitis With Polyposis
MeSH Terms: interventions — Budesonide; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- budesonide inhalation suspension (Experimental)
  Interventions: Drug: budesonide
- budesonide aqueous nasal spray (Active Comparator)
  Interventions: Drug: budesonide
- oral steroids (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: budesonide — 1mg/2ml Pulmicort Respules BIS twice daily
  Arms: budesonide inhalation suspension
Drug: budesonide — nasal spray 256μg BID
  Arms: budesonide aqueous nasal spray
Drug: Prednisone — oral prednisone 24mg QD
  Arms: oral steroids

SUMMARY:
Topical and systemic steroids constitute the first choice in medical treatment for nasal polyps. This study aimed to evaluate the efficacy and safety of a short course of budesonide inhalation suspension via transnasal nebulization in the preoperative management of chronic rhinosinusitis with nasal polyposis. The second aim was to compare budesonide inhalation suspension with budesonide aqueous nasal spray and oral prednisone in nasal polyp treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis was made on the basis of symptoms of rhinosinusitis (nasal obstruction, rhinorhea, loss of smell, and headache/facial pain) for at least 12 weeks, confirmed by abnormalities in all sinuses on computed tomography (CT) scan. The diagnosis of CRSwNP was based on the standard criteria issued in the European Position Paper on Rhinosinusitis and Nasal Polyps guidelines.
* Bilateral nasal polyps were present and endoscopic biopsy demonstrated eosinophilic polyposis. Patients were not recruited who had large polyps (total Kennedy score＝6).

Exclusion Criteria:

* a previous oral corticosteroid treatment.
* recent sinus surgery
* ASA intolerance
* cystic fibrosis
* pregnancy
* serious or unstable concurrent disease or psychological disorder.

Ages: 23 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-03 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical responses including 4 major symptoms(nasal obstruction, rhinorrhea, loss of smell,and headache/facial pain) | 2 weeks
  The primary efficacy outcome measure was the patients' assessment of four major symptoms improvement on an ordinal scaled visual analogue score of 0 to 10, where 0 indicates that no symptom is present and 10 signifies the presence of the most severe nasal obstruction, rhinorrhea, alteration in the sense of smell and headache/ facial pain.

SECONDARY OUTCOMES:
Physicians' assessment of nasal polyp size reduction | 2 weeks
  the physicians' assessment of nasal polyp size reduction by endoscopic examination according to Kennedy score (0, no polyps; 1, polyps in the middle meatus, not reaching below the inferior border of the middle turbinate; 2, polyps reaching below the inferior border of the middle turbinate, but not below the inferior border of the inferior turbinate; 3, large polyps reaching below the inferior turbinate). Bilateral polyp grade was obtained as the sum of the individual grades for the left and right nasal cavities. A total score of 0-6 is possible.